CLINICAL TRIAL: NCT04468100
Title: A Multicenter Prospective Randomized Comparative Study of Pharmacokinetics, Clinical Efficacy and Safety of Tigerase® (JSC GENERIUM, Russia) vs. Pulmozyme® (Hoffmann-La Roche, Switzerland) as Part of Complex Therapy in Patients With Cystic Fibrosis
Brief Title: Efficacy and Safety of Tigerase® vs. Pulmozyme® in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRN-CFR-III; 348 eff date 23.06.2017 (Other: Clinical trial approval number, Ministry of Health of Russia)
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis; Fibrosis
Keywords: Dornase; Cystic Fibrosis; Fibrosis; Lung Diseases; Pancreatic Diseases; Digestive System Diseases; Respiratory Tract Diseases; Pathologic Processes; Genetic Diseases, Inborn; Tigerase®; DNase
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis; Lung Diseases; Pancreatic Diseases; Digestive System Diseases; Respiratory Tract Diseases; Pathologic Processes; Genetic Diseases, Inborn | interventions — dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tigerase® (Experimental): Dornase alfa
  Interventions: Biological: Tigerase®
- Pulmozyme® (Active Comparator): Dornase alfa
  Interventions: Biological: Pulmozyme®

INTERVENTIONS:
Biological: Tigerase® — 2.5 mL (2.5 mg) dornase alfa nebulized once daily for 168 (+/-7) days
  Other Names: dornase alfa
  Arms: Tigerase®
Biological: Pulmozyme® — 2.5 mL (2.5 mg) dornase alfa nebulized once daily for 168 (+/-7) days
  Other Names: dornase alfa
  Arms: Pulmozyme®

SUMMARY:
It is a multicenter, open-label, randomized, parallel-group study of the efficacy and safety of Tigerase® compared Pulmozyme® in patients with Cystic Fibrosis

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a common hereditary disease with an autosomal recessive type of inheritance, characterized by systemic damage to the exocrine glands, mainly the bronchopulmonary and gastrointestinal systems. CF is usually characterized by a severe course and poor prognosis. The severity of the disease and the life expectancy of the patient with CF is determined primarily by the state of the bronchopulmonary system; more than 90% of patients die from lung diseases.

CF Pulmonary damage develops as a result of a gene mutation - cystic fibrosis transmembrane regulator of ion conductivity Na and Cl (CFTR-cystic fibrosis transmembrane regulator). The main function of CFTR is to regulate the transport of sodium and chlorine across the cell membrane and is part of the cAMP-dependent chlorine channel. CFTR-protein dysfunction in the bronchial tree epithelial cells leads to a blockage of the chlorine ions transport and an increase in the sodium ions absorption, and impaired fluid secretion through the epithelial cells apical membrane.

Dornase alpha, a human recombinant deoxyribonuclease 1 (rhDNase, rhDNase) hydrolyzes extracellular DNA (viscous polyanion) that enters the sputum from destroyed neutrophils, thereby reducing the adhesion and viscosity of sputum. In CF patients dornase alpha is used as symptomatic therapy in combination with standard therapy in patients with a forced vital capacity (FVC) index of at least 40% of the proper value.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Informed Consent Form for participation in the study;
2. Men and women 18 years and older;
3. Diagnosis of cystic fibrosis, defined as the presence of disease symptoms and a positive sweat test and / or detection of 2 mutations of the MVTR gene during genotyping;
4. FEV1 ≥40% and ≤100% of the proper value;
5. The ability to understand the protocol requirements, to give written consent to participate in the study (including the use and transfer of information about the patient's health status related to the study).

Exclusion Criteria:

1. Hypersensitivity to any of used study drug, to their components, as well as a history of significant allergic reactions;
2. Acute respiratory infection or exacerbation of chronic pulmonary disease within 4 weeks prior to screening and without corticosteroid or antibiotic therapy;
3. Concomitant diseases and conditions with potential impact the patients safety, including:

   * Severe renal impairment (serum creatinine more than 1.5 times higher than the upper limit of normal);
   * Severe liver impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) blood serum activity is 2.5 times or more higher than the upper limit of the laboratory norm);
4. A history of lung transplantation or planned transplantation during this study;
5. The presence of antibodies to HIV, active viral hepatitis B and / or C and / or cirrhosis in the history or detected on Screening;
6. Pregnancy and lactation;
7. Refusal of patients with preserved reproductive potential to use adequate contraception throughout the study and within 30 days after the end of the study;
8. Patients who underwent a blood or blood components transfusion within 10 days prior to screening;
9. Drug or alcohol abuse at the time of Screening or in the past;
10. Patient's participation in any other clinical trials and / or administration of an experimental drug within 30 days prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in the first second of a forced expiratory maneuver (FEV1) compared to baseline | FEV1 - forced expiratory volume in the first second of a forced expiratory maneuver by standard spirometry
  Week 24 ± 1

SECONDARY OUTCOMES:
Change in forced lung capacity (FVC) compared to baseline | Week 24 ± 1
  FVC - forced lung capacity by standard spirometry
The number of exacerbations of chronic pulmonary disease | Week 24 ± 1
  Clinical symptoms of chronic pulmonary disease exacerbation required antibiotic therapy in CF patients, include the presence of at least 4 of 12 possible signs or symptoms
  1. A change in color or amount of sputum;
  2. The appearance or intensification of hemoptysis;
  3. Strengthening cough;
  4. Increased shortness of breath;
  5. Increased malaise, fatigue or lethargy;
  6. Temperature above 38 ° C;
  7. Anorexia or weight loss;
  8. Sinuses pain or soreness;
  9. Changes in the nature of sinuses mucus;
  10. Changes in chest physical examination;
  11. Pulmonary function decrease at list 10% or more;
  12. Radiographic changes.
The number of days before the chronic pulmonary disease exacerbation development | Week 24 ± 1
Change in body weight compared to baseline | Week 24 ± 1
Change in the average score for the "Symptoms", "Activity", "Influence" subscales, as well as the average total score of the St. George's Respiratory Questionnaire (SGRQ), version 2.2 | Week 24 ± 1
  St. George's Respiratory Questionnaire (SGRQ), a questionnaire for patients with respiratory diseases is designed to assess the chronic obstructive pulmonary disease patients quality of life.
  The questionnaire consists of 76 questions, which are grouped in 3 parts:
  * The first part - symptoms - measures the degree of anxiety caused by respiratory symptoms.
  * The second part - activity - measures the limitation of mobility and physical activity.
  * The third part - the influence - evaluates the existing psychosocial consequences of bronchial obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (14):
- Russia (14):
  - Regional Clinical Hospital, Barnaul, Altayskiy Kray
  - Republican Clinical hospital named after G.G. Kuvatov, Ufa, Bashkortostan Republic
  - Crimean federal university named after V.I.Vernadsky, Simferopol, Crimea Republic
  - Sverdlovsk Regional clinical hospital No. 1, Yekaterinburg, Sverdlovsk Oblast
  - Kazan state medical University of Ministry of health, Hospital Therapy Department, Kazan', Tatarstan Republic
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - City Clinical Hospital named after D.D. Pletnev, Moscow
  - City Multidisciplinary Hospital No. 2, Saint Petersburg
  - Regional clinical Hospital, Saratov
  - Scientific medical center of General Medicine and pharmacologies, Stavropol
  - Tomsk national medical research Center of the Russian Academy of Sciences, Genetic Clinic Research Institute medical genetics, Tomsk
  - Volgograd State Medical University, Department of clinical pharmacology and intensive care, Volgograd
  - Children's Clinical Hospital No. 1 ", Cystic Fibrosis center, Yaroslavl
  - Clinical hospital No. 2, Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amelina EL, Krasovsky SA, Akhtyamova-Givirovskaya NE, Kashirskaya NY, Abdulganieva DI, Asherova IK, Zilber IE, Kozyreva LS, Kudelya LM, Ponomareva ND, Revel-Muroz NP, Reutskaya EM, Stepanenko TA, Seitova GN, Ukhanova OP, Magnitskaya OV, Kudlay DA, Markova OA, Gapchenko EV. Comparison of biosimilar Tigerase and Pulmozyme in long-term symptomatic therapy of patients with cystic fibrosis and severe pulmonary impairment (subgroup analysis of a Phase III randomized open-label clinical trial (NCT04468100)). PLoS One. 2021 Dec 23;16(12):e0261410. doi: 10.1371/journal.pone.0261410. eCollection 2021. PMID 34941914
- See also: Efficacy and safety of the biosimilar medicinal product Tigerase® (dornase alfa) in long-term symptomatic treatment of patients with cystic fibrosis: results of a phase III clinical trial — https://www.researchgate.net/publication/339557202_Efficacy_and_safety_of_the_biosimilar_medicinal_product_TigeraseR_dornase_alfa_in_long-term_symptomatic_treatment_of_patients_with_cystic_fibrosis_results_of_a_phase_III_clinical_trial